CLINICAL TRIAL: NCT00002006
Title: A Phase I/II Pilot Study of Simultaneously Administered Rhu GM-CSF ( CHO Cell ) and Azidothymidine ( AZT ) in Patients With Severe HIV Infection and Leukopenia: Pharmacokinetics and Feasibility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 067A; 07936
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-01

CONDITIONS: HIV Infections; Cytopenias
Keywords: Neutropenia; Drug Interactions; Granulocyte-Macrophage Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Cytopenia; Neutropenia; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; sargramostim

INTERVENTIONS:
Drug: Zidovudine
Drug: Sargramostim

SUMMARY:
To assess the safety and efficacy of subcutaneously administered sargramostim ( granulocyte-macrophage colony-stimulating factor; GM-CSF ) in increasing and maintaining the neutrophil count in HIV-infected adults who have developed neutropenia as a result of receiving the antiretroviral agent, zidovudine ( AZT ). To assess the safety and efficacy of subcutaneously administered GM-CSF in increasing and maintaining the neutrophil count in HIV-infected adults with pre-existing neutropenia who are at high risk of developing hematologic intolerance while receiving the antiretroviral agent, AZT, for the first time. To assess the potential therapeutic benefit of concomitant GM-CSF and AZT on the natural history of HIV infection and associated infectious complications.

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed:

* Minimal local irradiation for tumors.

Patients must have:

* Diagnosis of AIDS or AIDS related complex (ARC).
* Neutropenia, due either to zidovudine (AZT) or HIV infection.
* Life expectancy = or > 6 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Significant malabsorption as defined by greater than 10 percent weight loss and one or more of the following:
* Serum carotene less than 75 IU/ml.
* Vitamin A level less than 75 IU/ml.
* More than 4 foul-smelling or greasy stools per day.
* Other criteria of malabsorption.
* Kaposi's sarcoma (KS) or other tumor which is likely to require specific antitumor therapy during study, other than minimal local irradiation.
* Active, life-threatening infection with bacterial, viral, fungal, or protozoan pathogens or fever of 39 degrees C within 10 days of study entry, unless it is apparent that the fever is not due to a severe underlying infection.

Concurrent Medication:

Excluded within 4 weeks of study entry:

* Any investigational drug.
* Immunomodulating agents.
* Hormonal therapy.
* Cytolytic chemotherapeutic agents.
* Antiretroviral agent other than zidovudine (AZT).
* Excluded within 4 months of study entry:
* Suramin.
* Excluded within 3 months of study entry:
* Ribavirin.

Patients with the following are excluded:

* Significant malabsorption.
* Tumor likely to require specific antitumor therapy during study.
* Other significant medical problems and conditions specified in Patient Exclusion Co-Existing Conditions.
* Uncorrected nutritional deficiencies that may contribute to neutropenia.
* Hypersensitivity to zidovudine (AZT) or other nucleoside analogs.
* Profound dementia or altered mental status that would prohibit the giving of informed consent.

Prior Treatment:

Excluded within 1 month of study entry:

* Transfusion.
* Excluded within 4 weeks of study entry:
* Radiation therapy to greater than 100 cm2 body area.

Current drug or alcohol abuse. Unprotected sexual behavior or other activities which might introduce a new inoculation of HIV during the study.

Patients must be willing to refrain from unprotected sexual or other activities which might introduce a new inoculum of HIV during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Natl Cancer Institute, Bethesda, Maryland, United States

REFERENCES:
- [Background] Levine JD, Allan JD, Tessitore JH, Falcone N, Galasso F, Israel RJ, Groopman JE. Recombinant human granulocyte-macrophage colony-stimulating factor ameliorates zidovudine-induced neutropenia in patients with acquired immunodeficiency syndrome (AIDS)/AIDS-related complex. Blood. 1991 Dec 15;78(12):3148-54. PMID 1742482